CLINICAL TRIAL: NCT01460186
Title: Evaluation of the Predictive and Prognostic Value of Germ-line Polymorphisms in Patients With Metastatic Breast Cancer : a Multicenter Non-randomized Prospective Cohort Study
Brief Title: Evaluation of the Predictive and Prognostic Value of Germ-line Polymorphisms in Patients With Metastatic Breast Cancer
Acronym: StoRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Centre de Recherche en Cancérologie de Lyon (Unknown)
Responsible Party: Sponsor
Purpose: Other
Other Study IDs: StoRM
Record Dates: First submitted 2011-08-02; First posted 2011-10-26 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Metastasis
Keywords: Germ line polymorphisms
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood samples (Experimental)
  Interventions: Other: Blood sample for genetic analysis (Identification of germ line genetic factors that influence the risk of metastatic breast cancer)

INTERVENTIONS:
Other: Blood sample for genetic analysis (Identification of germ line genetic factors that influence the risk of metastatic breast cancer) — Blood samples will be collected in one 6 ml EDTA and one 6 ml ACD tube after informed consent and inclusion in the study.

SUMMARY:
This is a multicenter, non-randomized, prospective cohort study. The purpose of the study is to identify germ line genetic factors that influence the risk of metastatic breast cancer.

1500 patients will be enrolled in this study. Blood samples will be collected after informed consent and inclusion in the study.

Patients will be treated and followed according to the standards of their treating center.

They will be followed during at least 5 years every 6 months for 3 years then every year.

DETAILED DESCRIPTION:
The StoRM trial is designed for analysis in association with the SIGNAL study which aims to decipher the genetic risk of breast cancer displaying amplification of the HER2 gene as well as resistance or toxicity to adjuvant treatments. SIGNAL study is in the process of recruiting 6000 localized breast cancer patients.

The purpose of the StoRM trial is to create a cohort of 1500 patients with metastatic breast cancer including detailed epidemiologic and treatment data. Using germ line polymorphisms in these patients and comparing them to patients with localized cancer from the SIGNAL study, the investigators will answer questions specific to the genetic influence on the prognosis of breast cancer and its response to treatments in the metastatic phase.

Blood samples will be collected in one 6 ml EDTA and one 6 ml ACD tube after informed consent and inclusion in the study. To simplify the evolution of the study and to avoid all confusion, the sample collection procedures followed will be identical to those used in the SIGNAL study.

As the samples are received at the biological resource center, the plasma will be aliquoted into a 500 µl tube and frozen at -80° C. DNA will be extracted using standard protocols. Plasma and DNA will be stored in anticipation of genetic analyses. An aliquot of the DNA sample will be genotyped for a panel of high-density genetic markers covering the whole genome, for genome-wide association studies.

The collected plasma may also be used for analyses to determine the expression profile of proteins, alone or combined with genetic factors that allow distinguishing between groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with a histologically proven breast adenocarcinoma, with metastatic progression diagnosed within one year (inclusion of patients who have a metastatic progression more than one year ago would favor the inclusion of patients with indolent cancer, possibly biasing the study) or locally advanced (no curative treatment)
* ER, PR and HER2 status known
* Age >= 18 years
* Affiliation with a social security scheme
* Signed informed consent

Exclusion Criteria:

* Coexisting or other cancer diagnosed within the previous 5 years that may be responsible for the current metastasis
* Patient who cannot follow medical surveillance due to geographical, social or psychological reasons
* Patient included in the SIGNAL study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2011-12 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Germ line genetic factors associated with metastatic relapse | at the end of enrollment (2 years)
  Genetic determinants that predispose to a metastatic relapse of brest cancer by establishing germ line genetic variation based on single nucleotide polymorphisms of patients with metastatic breast cancer and comparing this variation to a cohort of patients with localized breast cancer (SIGNAL study)(correlation between polymorphisms and risk of relapse)

SECONDARY OUTCOMES:
Genetic determinants that predispose to specific metastatic localizations | at the end of enrollment (2 years)
  Germ line polymorphisms will be analysed and tested for association with specific metastatic localizations as bone, lung, liver or central nervous system.
Genetic determinants that predispose to metastatic relapse of specific molecular subtype of breast cancer | at the end of enrollment (2 years)
  Germ line polymorphisms will be analysed and tested for association with metastatic relapse as a function of immunohistochemical/molecular characteristics of the primary tumor
Overall survival | At the end of the study (7 years: 2 years of enrollment and 5 years of follow-up)
  Evaluate as a function of germ line polymorphisms overall survival after first-line treatment in metastatic setting
Progression free survival | At the end of the study (7 years: 2 years of enrollment and 5 years of follow-up)
  Evaluate as a function of germ line polymorphisms progression free survival after first-line treatment in metastatic setting

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BACHELOT, MD, Principal Investigator — Centre Leon Berard
Locations (17):
- France (17):
  - Hôpital Jean Minjoz - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Institut Daniel Hollard, Grenoble
  - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Sainsbury JR, Anderson TJ, Morgan DA, Dixon JM. ABC of breast diseases. Breast cancer. BMJ. 1994 Oct 29;309(6962):1150-3. doi: 10.1136/bmj.309.6962.1150. No abstract available. PMID 7755703
- [Background] Vargo-Gogola T, Rosen JM. Modelling breast cancer: one size does not fit all. Nat Rev Cancer. 2007 Sep;7(9):659-72. doi: 10.1038/nrc2193. PMID 17721431
- [Background] Ansieau S, Bastid J, Doreau A, Morel AP, Bouchet BP, Thomas C, Fauvet F, Puisieux I, Doglioni C, Piccinin S, Maestro R, Voeltzel T, Selmi A, Valsesia-Wittmann S, Caron de Fromentel C, Puisieux A. Induction of EMT by twist proteins as a collateral effect of tumor-promoting inactivation of premature senescence. Cancer Cell. 2008 Jul 8;14(1):79-89. doi: 10.1016/j.ccr.2008.06.005. PMID 18598946
- [Background] Ramshaw IA, Carlsen S, Wang HC, Badenoch-Jones P. The use of cell fusion to analyse factors involved in tumour cell metastasis. Int J Cancer. 1983 Oct 15;32(4):471-8. doi: 10.1002/ijc.2910320414. PMID 6684641
- [Background] Tuck AB, Wilson SM, Chambers AF. ras transfection and expression does not induce progression from tumorigenicity to metastatic ability in mouse LTA cells. Clin Exp Metastasis. 1990 Sep-Oct;8(5):417-31. doi: 10.1007/BF00058153. PMID 1697227
- [Background] Lifsted T, Le Voyer T, Williams M, Muller W, Klein-Szanto A, Buetow KH, Hunter KW. Identification of inbred mouse strains harboring genetic modifiers of mammary tumor age of onset and metastatic progression. Int J Cancer. 1998 Aug 12;77(4):640-4. doi: 10.1002/(sici)1097-0215(19980812)77:43.0.co;2-8. PMID 9679770
- [Background] Udler M, Pharoah PD. Germline genetic variation and breast cancer survival: prognostic and therapeutic implications. Future Oncol. 2007 Oct;3(5):491-5. doi: 10.2217/14796694.3.5.491. No abstract available. PMID 17927512
- [Background] Hemminki K, Ji J, Forsti A, Sundquist J, Lenner P. Survival in breast cancer is familial. Breast Cancer Res Treat. 2008 Jul;110(1):177-82. doi: 10.1007/s10549-007-9692-7. Epub 2007 Aug 3. PMID 17674192
- [Background] Cox A, Dunning AM, Garcia-Closas M, Balasubramanian S, Reed MW, Pooley KA, Scollen S, Baynes C, Ponder BA, Chanock S, Lissowska J, Brinton L, Peplonska B, Southey MC, Hopper JL, McCredie MR, Giles GG, Fletcher O, Johnson N, dos Santos Silva I, Gibson L, Bojesen SE, Nordestgaard BG, Axelsson CK, Torres D, Hamann U, Justenhoven C, Brauch H, Chang-Claude J, Kropp S, Risch A, Wang-Gohrke S, Schurmann P, Bogdanova N, Dork T, Fagerholm R, Aaltonen K, Blomqvist C, Nevanlinna H, Seal S, Renwick A, Stratton MR, Rahman N, Sangrajrang S, Hughes D, Odefrey F, Brennan P, Spurdle AB, Chenevix-Trench G; Kathleen Cunningham Foundation Consortium for Research into Familial Breast Cancer; Beesley J, Mannermaa A, Hartikainen J, Kataja V, Kosma VM, Couch FJ, Olson JE, Goode EL, Broeks A, Schmidt MK, Hogervorst FB, Van't Veer LJ, Kang D, Yoo KY, Noh DY, Ahn SH, Wedren S, Hall P, Low YL, Liu J, Milne RL, Ribas G, Gonzalez-Neira A, Benitez J, Sigurdson AJ, Stredrick DL, Alexander BH, Struewing JP, Pharoah PD, Easton DF; Breast Cancer Association Consortium. A common coding variant in CASP8 is associated with breast cancer risk. Nat Genet. 2007 Mar;39(3):352-8. doi: 10.1038/ng1981. Epub 2007 Feb 11. PMID 17293864
- [Background] Thomas G, Jacobs KB, Kraft P, Yeager M, Wacholder S, Cox DG, Hankinson SE, Hutchinson A, Wang Z, Yu K, Chatterjee N, Garcia-Closas M, Gonzalez-Bosquet J, Prokunina-Olsson L, Orr N, Willett WC, Colditz GA, Ziegler RG, Berg CD, Buys SS, McCarty CA, Feigelson HS, Calle EE, Thun MJ, Diver R, Prentice R, Jackson R, Kooperberg C, Chlebowski R, Lissowska J, Peplonska B, Brinton LA, Sigurdson A, Doody M, Bhatti P, Alexander BH, Buring J, Lee IM, Vatten LJ, Hveem K, Kumle M, Hayes RB, Tucker M, Gerhard DS, Fraumeni JF Jr, Hoover RN, Chanock SJ, Hunter DJ. A multistage genome-wide association study in breast cancer identifies two new risk alleles at 1p11.2 and 14q24.1 (RAD51L1). Nat Genet. 2009 May;41(5):579-84. doi: 10.1038/ng.353. Epub 2009 Mar 29. PMID 19330030
- [Background] Lander ES, Linton LM, Birren B, Nusbaum C, Zody MC, Baldwin J, Devon K, Dewar K, Doyle M, FitzHugh W, Funke R, Gage D, Harris K, Heaford A, Howland J, Kann L, Lehoczky J, LeVine R, McEwan P, McKernan K, Meldrim J, Mesirov JP, Miranda C, Morris W, Naylor J, Raymond C, Rosetti M, Santos R, Sheridan A, Sougnez C, Stange-Thomann Y, Stojanovic N, Subramanian A, Wyman D, Rogers J, Sulston J, Ainscough R, Beck S, Bentley D, Burton J, Clee C, Carter N, Coulson A, Deadman R, Deloukas P, Dunham A, Dunham I, Durbin R, French L, Grafham D, Gregory S, Hubbard T, Humphray S, Hunt A, Jones M, Lloyd C, McMurray A, Matthews L, Mercer S, Milne S, Mullikin JC, Mungall A, Plumb R, Ross M, Shownkeen R, Sims S, Waterston RH, Wilson RK, Hillier LW, McPherson JD, Marra MA, Mardis ER, Fulton LA, Chinwalla AT, Pepin KH, Gish WR, Chissoe SL, Wendl MC, Delehaunty KD, Miner TL, Delehaunty A, Kramer JB, Cook LL, Fulton RS, Johnson DL, Minx PJ, Clifton SW, Hawkins T, Branscomb E, Predki P, Richardson P, Wenning S, Slezak T, Doggett N, Cheng JF, Olsen A, Lucas S, Elkin C, Uberbacher E, Frazier M, Gibbs RA, Muzny DM, Scherer SE, Bouck JB, Sodergren EJ, Worley KC, Rives CM, Gorrell JH, Metzker ML, Naylor SL, Kucherlapati RS, Nelson DL, Weinstock GM, Sakaki Y, Fujiyama A, Hattori M, Yada T, Toyoda A, Itoh T, Kawagoe C, Watanabe H, Totoki Y, Taylor T, Weissenbach J, Heilig R, Saurin W, Artiguenave F, Brottier P, Bruls T, Pelletier E, Robert C, Wincker P, Smith DR, Doucette-Stamm L, Rubenfield M, Weinstock K, Lee HM, Dubois J, Rosenthal A, Platzer M, Nyakatura G, Taudien S, Rump A, Yang H, Yu J, Wang J, Huang G, Gu J, Hood L, Rowen L, Madan A, Qin S, Davis RW, Federspiel NA, Abola AP, Proctor MJ, Myers RM, Schmutz J, Dickson M, Grimwood J, Cox DR, Olson MV, Kaul R, Raymond C, Shimizu N, Kawasaki K, Minoshima S, Evans GA, Athanasiou M, Schultz R, Roe BA, Chen F, Pan H, Ramser J, Lehrach H, Reinhardt R, McCombie WR, de la Bastide M, Dedhia N, Blocker H, Hornischer K, Nordsiek G, Agarwala R, Aravind L, Bailey JA, Bateman A, Batzoglou S, Birney E, Bork P, Brown DG, Burge CB, Cerutti L, Chen HC, Church D, Clamp M, Copley RR, Doerks T, Eddy SR, Eichler EE, Furey TS, Galagan J, Gilbert JG, Harmon C, Hayashizaki Y, Haussler D, Hermjakob H, Hokamp K, Jang W, Johnson LS, Jones TA, Kasif S, Kaspryzk A, Kennedy S, Kent WJ, Kitts P, Koonin EV, Korf I, Kulp D, Lancet D, Lowe TM, McLysaght A, Mikkelsen T, Moran JV, Mulder N, Pollara VJ, Ponting CP, Schuler G, Schultz J, Slater G, Smit AF, Stupka E, Szustakowki J, Thierry-Mieg D, Thierry-Mieg J, Wagner L, Wallis J, Wheeler R, Williams A, Wolf YI, Wolfe KH, Yang SP, Yeh RF, Collins F, Guyer MS, Peterson J, Felsenfeld A, Wetterstrand KA, Patrinos A, Morgan MJ, de Jong P, Catanese JJ, Osoegawa K, Shizuya H, Choi S, Chen YJ, Szustakowki J; International Human Genome Sequencing Consortium. Initial sequencing and analysis of the human genome. Nature. 2001 Feb 15;409(6822):860-921. doi: 10.1038/35057062. PMID 11237011
- [Background] Olivier M, Aggarwal A, Allen J, Almendras AA, Bajorek ES, Beasley EM, Brady SD, Bushard JM, Bustos VI, Chu A, Chung TR, De Witte A, Denys ME, Dominguez R, Fang NY, Foster BD, Freudenberg RW, Hadley D, Hamilton LR, Jeffrey TJ, Kelly L, Lazzeroni L, Levy MR, Lewis SC, Liu X, Lopez FJ, Louie B, Marquis JP, Martinez RA, Matsuura MK, Misherghi NS, Norton JA, Olshen A, Perkins SM, Perou AJ, Piercy C, Piercy M, Qin F, Reif T, Sheppard K, Shokoohi V, Smick GA, Sun WL, Stewart EA, Fernando J, Tejeda, Tran NM, Trejo T, Vo NT, Yan SC, Zierten DL, Zhao S, Sachidanandam R, Trask BJ, Myers RM, Cox DR. A high-resolution radiation hybrid map of the human genome draft sequence. Science. 2001 Feb 16;291(5507):1298-302. doi: 10.1126/science.1057437. PMID 11181994
- [Background] Azzato EM, Pharoah PD, Harrington P, Easton DF, Greenberg D, Caporaso NE, Chanock SJ, Hoover RN, Thomas G, Hunter DJ, Kraft P. A genome-wide association study of prognosis in breast cancer. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1140-3. doi: 10.1158/1055-9965.EPI-10-0085. Epub 2010 Mar 23. PMID 20332263
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901